CLINICAL TRIAL: NCT05934617
Title: Trajectories of FEV1 After Lung Transplantation: Determinants and Clinical Outcomes
Brief Title: Trajectories of FEV1 After Lung Transplantation
Acronym: TRAJLUNG
Status: Enrolling by invitation | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: TRAJLUNG001
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Lung Transplant Failure and Rejection; Chronic Lung Allograft Dysfunction
Keywords: Lung trajectories; Unsupervised analysis; Determinants of FEV1 trajectories
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Foch hospital: Lung recipients from Foch hospital, Suresnes, France
- Bichat hospital: Lung recipients from Bichat hospital, Paris, France
- Nantes hospital: Lung recipients from Nantes hospital, Nantes, France
- San Antonio center: Lung recipients from Pulmonary hypertension center, San Antonio, Texas, US
- Marie-Lannelongue hospital: Lung recipients from Marie-Lannelongue hospital, Le Plessis-Robinson, France
- Bordeaux hospital: Lung recipients from Bordeaux hospital, Nantes, France
- Marseille hospital: Lung recipients from Marseille hospital, Marseille, France
- Toulouse hospital: Lung recipients from Toulouse hospital, Toulouse, France
- Strasbourg hospital: Lung recipients from Strasbourg hospital, Strasbourg, France
- Grenoble hospital: Lung recipients from Grenoble hospital, Grenoble, France
- Cochin hospital: Lung recipients from Strasbourg hospital, Paris, France
- Hospital center Mayenne North: Lung recipients from Hospital center Mayenne North, Mayenne, France

SUMMARY:
For individuals with ESLD, lung transplantation is the best, or only treatment option with increased pulmonary function and quality of life. The forced expiratory volume in one second (FEV1) is the standard to monitor the lung function after transplantation. The goal of this study is to identify and validate the FEV1 trajectories after lung transplantation, as well as their determinants and outcomes, using an international cohort of lung recipients.

DETAILED DESCRIPTION:
Chronic lung diseases affect about 500 million individuals and are the third leading cause of death worldwide, accounting for 7% of all mortality. They drive the growing number of individuals with end stage lung disease (ESLD), a public health issue with socioeconomic consequences.

For individuals with ESLD, lung transplantation is the best, or only treatment option with increased pulmonary function and quality of life. Lung recipients remain however particularly at risk, with a median patient survival of around five years, which is much lower than other organ recipients, such as kidney, heart or liver recipients. Adequate monitoring of the lung recipient is therefore crucial to optimize the allograft longevity.

The forced expiratory volume in one second (FEV1) is the standard to monitor the lung function after transplantation, and is used to evaluate the stage and severity of lung allograft diseases. However, according to a literature review we performed, the very few studies that have investigated the FEV1 evolution, and its relationship with outcomes such as death or chronic lung allograft dysfunction, were commonly based on cohort with insufficient data variety and completeness. Importantly, these studies lacked external validation, multidimensional approach, and none has attempted to identify the main profiles of FEV1 trajectories and their associated parameters. As such, the determinants and long-term outcomes of FEV1 trajectories are still poorly understood.

A multidimensional, trajectory-based approach may help unveil clinically relevant organ function profiles among lung recipients. Indeed, several studies have shown the potential existence of underlying trajectories of transplanted organs' function and diseases, and their associations with outcomes and relevance for patient management, such as in kidney or heart transplantation. These studies used a unsupervised approach, which permitted to erase any preconceived clinical ideas. Overall, this approach has shown its value in several medical specialties, in particular in image analysis, oncology, or cardiology.

Therefore, the goal of this study was to identify and validate the FEV1 trajectories after lung transplantation, as well as their determinants and outcomes, using an international cohort of lung recipients, with a protocol-based collection of FEV1 repeated assessments and clinical, biological, histological and immunological data.

ELIGIBILITY:
Inclusion Criteria:

* Double lung transplant recipients
* Age 18 years or older at the time of transplant
* Transplant between January 1, 2010 and December 31, 2020
* At least 2 PFTs available for analysis

Exclusion Criteria:

* Did not consent to clinical data use for research purposes
* Multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who received a bilateral lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
FEV1 trajectories | Up to 10 years after lung transplantation
  FEV1 trajectories of the lung recipient

SECONDARY OUTCOMES:
Patient death | Up to 10 years after lung transplantation
  Patient death after lung transplantation
Allograft failure | Up to 10 years after lung transplantation
  Allograft failure after lung transplantation
Chronic lung allograft dysfunction | Up to 10 years after lung transplantation
  CLAD after lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Roux, MD, PhD, Principal Investigator — Foch hospital
Locations (1):
- Foch hospital, Suresnes, France

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data may be shared for research purpose upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: Via email to the corresponding author

REFERENCES:
- [Background] GBD Chronic Respiratory Disease Collaborators. Prevalence and attributable health burden of chronic respiratory diseases, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Respir Med. 2020 Jun;8(6):585-596. doi: 10.1016/S2213-2600(20)30105-3. PMID 32526187
- [Background] Li X, Cao X, Guo M, Xie M, Liu X. Trends and risk factors of mortality and disability adjusted life years for chronic respiratory diseases from 1990 to 2017: systematic analysis for the Global Burden of Disease Study 2017. BMJ. 2020 Feb 19;368:m234. doi: 10.1136/bmj.m234. PMID 32075787
- [Background] Brakema EA, Tabyshova A, van der Kleij RMJJ, Sooronbaev T, Lionis C, Anastasaki M, An PL, Nguyen LT, Kirenga B, Walusimbi S, Postma MJ, Chavannes NH, van Boven JFM; FRESH AIR collaborators. The socioeconomic burden of chronic lung disease in low-resource settings across the globe - an observational FRESH AIR study. Respir Res. 2019 Dec 21;20(1):291. doi: 10.1186/s12931-019-1255-z. PMID 31864411
- [Background] Perch M, Hayes D Jr, Cherikh WS, Zuckermann A, Harhay MO, Hsich E, Potena L, Sadavarte A, Lindblad K, Singh TP, Stehlik J; International Society for Heart and Lung Transplantation. The International Thoracic Organ Transplant Registry of the International Society for Heart and Lung Transplantation: Thirty-ninth adult lung transplantation report-2022; focus on lung transplant recipients with chronic obstructive pulmonary disease. J Heart Lung Transplant. 2022 Oct;41(10):1335-1347. doi: 10.1016/j.healun.2022.08.007. Epub 2022 Aug 20. No abstract available. PMID 36050206